CLINICAL TRIAL: NCT04389450
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel-Group Phase II Study to Evaluate the Efficacy and Safety of Intramuscular Injections of PLX PAD for the Treatment of Severe COVID-19
Brief Title: Double-Blind, Multicenter, Study to Evaluate the Efficacy of PLX PAD for the Treatment of COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The decision to bring the Study to early clinical readout came in response to COVID-19's evolution as a disease, and the significant changes in the standard of care, leading to an increase in the severity of conditions of the intubated patients
Sponsor: Pluristem Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PLX-COV-01
Record Dates: First submitted 2020-05-14; First posted 2020-05-15 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: COVID; ARDS

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- PLX-PAD interval high dose (Experimental): PLX-PAD will be administered via 15 IM injections (1 mL each). Each subject will be treated twice, with an interval of 1 week between treatments.
  Interventions: Biological: PLX-PAD
- PLX-PAD low dose (Experimental): PLX-PAD 300, single administration, second administration of placebo after 1 week.
  Interventions: Biological: PLX-PAD
- Control Group A (Placebo Comparator): Placebo, two administrations, 1 week apart
  Interventions: Biological: Placebo
- PLX-PAD high dose (Experimental): PLX-PAD, single administration
  Interventions: Biological: PLX-PAD
- Control Group B (Placebo Comparator): Placebo, single administration
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: PLX-PAD — PLX-PAD, allogeneic ex vivo expanded placental mesenchymal-like adherent stromal cells
  Arms: PLX-PAD high dose; PLX-PAD interval high dose; PLX-PAD low dose
Biological: Placebo — Placebo solution for injection
  Arms: Control Group A; Control Group B

SUMMARY:
This clinical trial will examine if a new treatment of Mesenchymal-like Adherent stromal Cells (called PLX-PAD) can help patients intubated and mechanically ventilated due to COVID-19 to recover more quickly with less complications.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent, or with a legal representative who can provide informed consent.
* Male or non-pregnant female adult 40-80 years of age at time of enrollment.
* Laboratory-confirmed SARS-CoV-2 infection as determined by PCR, in any specimen up to 21 days prior to randomization.
* Meets definition of ARDS according to Berlin criteria.

Key Exclusion Criteria:

* Body weight under 55 kg (121 lbs)
* Serum creatinine level of over 1.5 mg/dL at time of randomization.
* Total Bilirubin ≥2 mg/dL at time of randomization.
* Known allergy to any of the following: dimethyl sulfoxide (DMSO), human serum albumin, bovine serum albumin.
* Stroke or acute myocardial infarction/unstable angina within 3 months prior to randomization.
* Chronic Obstructive Pulmonary disease GOLD stage above II.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Number of ventilator free days | 28 days

SECONDARY OUTCOMES:
All-cause mortality | 28 days
Duration of mechanical ventilation | 8 weeks

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - University of California Irvine, Irvine, California
  - University of Southern California (USC) - Keck School of Medicine (KSOM), Los Angeles, California
  - University Of California Davis,4860 Y Street, Sacramento, California
  - Baptist Health Medical Center, Jacksonville, Florida
  - Medical College of Georgia at Augusta University, Augusta, Georgia
  - Sarah Cannon Research Institute, LLC (Mercer University School of Medicine), Macon, Georgia
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cooper Research Institute, Camden, New Jersey
  - Holy Medical Center, Teaneck, New Jersey
  - Montefiore Medical Center, New York, New York
  - Maimonides Medical Center, New York, New York
  - Mercy Medical Center, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.pluristem.com